CLINICAL TRIAL: NCT04213924
Title: The Analgesic Efficacy of Ultrasound-Guided Erector Spinae Plan Block in Patients Undergoing ESWL
Brief Title: Ultrasound-Guided Erector Spinae Plan Block in Patients Undergoing ESWL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ahmet Murat Yayik, Assistant Professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ESPB for ESWL
Record Dates: First submitted 2019-12-27; First posted 2019-12-30 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Urinary System Stones; Pain
Keywords: Extracorporeal Shockwave Lithotripsy; Erector Spinae Plane Block
MeSH Terms: conditions — Pain | interventions — Bupivacaine; Lidocaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group ESPB (Active Comparator): Ultrasound-guided erector spinae plane block with 10 ml %0.5 bupivacaine and 10 ml %2 lidocaine
  Interventions: Drug: Bupivacaine HCl 0.5 % in 10 ml and 2 % lidocaine in 10 ml
- Group NSAII (Active Comparator): lidocaine 5% gel and 800 mg ibuprofen intravenously
  Interventions: Drug: 5 % Lidocaine Topical Gel and 800 mg ibuprofen intravenously

INTERVENTIONS:
Drug: Bupivacaine HCl 0.5 % in 10 ml and 2 % lidocaine in 10 ml — Erector spinae plane block, 30 min before the ESWL procedure.
  Arms: Group ESPB
Drug: 5 % Lidocaine Topical Gel and 800 mg ibuprofen intravenously — 5 % Lidocaine Topical Gel and 800 mg ibuprofen intravenously, 30 min before the ESWL procedure.
  Arms: Group NSAII

SUMMARY:
Extracorporeal shock wave lithotripsy (ESWL) is widely used in the treatment of urinary tract stones and is generally applied to outpatients. To achieve fragmentation in ESWL, shock waves must be applied with sufficient power and time. Providing effective analgesia during this procedure is crucial to the success of the procedure. Erector Spinae Plan Block (ESPB) was first described in 2016 and, it is frequently used for postoperative analgesia in urinary system surgery. This study aimed to investigate the efficacy of ESPB in patients undergoing ESWL.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist's physiologic state I-II patients undergoing Extracorporeal Shockwave Lithotripsy

Exclusion Criteria:

* chronic pain
* bleeding disorders
* renal or hepatic insufficiency
* patients on chronic non-steroidal anti-inflammatory medications
* emergency cases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Opioid Consumption | Intraoperative 30 minutes
  Opioid consumption during procedure

SECONDARY OUTCOMES:
Visual Analog Pain Score | Intraoperative 30 minutes
  Pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

REFERENCES:
- [Background] Yayik AM, Ahiskalioglu A, Alici HA, Celik EC, Cesur S, Ahiskalioglu EO, Demirdogen SO, Karaca O, Adanur S. Less painful ESWL with ultrasound-guided quadratus lumborum block: a prospective randomized controlled study. Scand J Urol. 2019 Dec;53(6):411-416. doi: 10.1080/21681805.2019.1658636. Epub 2019 Sep 9. PMID 31496381
- [Background] Yayik AM, Celik EC, Ahiskalioglu A. An unusual usage for ultrasound guided Quadratus Lumborum Block: Pediatric extracorporeal shock wave lithotripsy. J Clin Anesth. 2018 May;46:47-48. doi: 10.1016/j.jclinane.2018.01.016. Epub 2018 Mar 26. No abstract available. PMID 29414615